CLINICAL TRIAL: NCT01109316
Title: An Open-Label, Randomized, Crossover Trial of CSII Reservoir In-use Comparing Insulin Lispro Formulation to Insulin Aspart in Patients With Type 1 Diabetes Mellitus
Brief Title: Insulin Lispro 6 Days Versus Insulin Aspart 6 Days in Pump Use
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 12174; F3Z-MC-IOPV (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-04-19; First posted 2010-04-23 (Estimated); Results first posted 2012-10-30 (Estimated); Last update posted 2019-03-27 (Actual); Status verified 2019-03

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Lispro; Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Insulin Lispro 2 Day (Active Comparator)
  Interventions: Drug: Insulin lispro 2 day reservoir in-use
- Insulin Lispro 6 Day (Experimental)
  Interventions: Drug: Insulin lispro 6 day reservoir in-use
- Insulin Aspart 6 Day (Active Comparator)
  Interventions: Drug: Insulin aspart 6 day reservoir in-use

INTERVENTIONS:
Drug: Insulin lispro 2 day reservoir in-use — Insulin lispro 2 Day (L2D) administered by infusion pump for 8 week treatment period.
  Other Names: LY275585; Humalog
  Arms: Insulin Lispro 2 Day
Drug: Insulin lispro 6 day reservoir in-use — Insulin lispro 6 Day (L6D) administered by infusion pump for 8 week treatment period.
  Other Names: LY275585; Humalog
  Arms: Insulin Lispro 6 Day
Drug: Insulin aspart 6 day reservoir in-use — Insulin aspart 6 Day (A6D) administered by infusion pump for 8 week treatment period.
  Arms: Insulin Aspart 6 Day

SUMMARY:
This is a 6-sequence, 3-period (8 weeks each), 3-arm, 24-week crossover study. The purpose of this study is to provide information on the use of insulin lispro in insulin pumps (Continuous Subcutaneous Insulin Infusion [CSII]) compared to insulin aspart over 6 days of pump reservoir in-use. The study will also compare the in-use characteristics of insulin lispro infused at 6 days with insulin lispro infused at 2 days.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 1 diabetes (World Health Organization criteria) for at least 24 months.
* Treated with continuous subcutaneous insulin infusion therapy for the previous 6 months.
* Mean total daily insulin dose for 3 days prior to screening equal to or less than 46 units/day using a 300-unit reservoir or less than or equal to 26 units/day using a 180 unit reservoir.
* Baseline body mass index (BMI) less than or equal to 35.0 kg/m^2.
* Baseline glycosylated hemoglobin (HbA1c) 5% to 9%.

Exclusion Criteria:

* Impaired renal function (serum creatinine greater than or equal to 2.0 milligrams per deciliter [mg/dL]).
* Legal blindness.
* Have had any episode of hypoglycemic coma, seizures, or disorientation in the 12 months prior to screening.
* Have had hypoglycemia unawareness (routinely asymptomatic at blood glucose (BG) less than 45 mg/dL) in the 12 months prior to screening.
* Have had any emergency room visits or hospitalizations due to poor glucose control in the 12 months prior to screening.
* Have had a pump-related infusion site abscess in the 12 months prior to screening.
* Have had multiple, clinically significant occlusions as judged by the investigator.
* Have had any infection with staphylococcus aureus in the past 5 years.
* Have one of the following concomitant diseases: presence of clinically significant hematologic, oncologic, renal, cardiac, hepatic, or gastrointestinal disease, or any other serious disease considered by the investigator to be exclusionary.
* Patients with malignancy other than basal cell or squamous cell skin cancer who have not yet been treated, are currently being treated, or who were diagnosed less than 5 years ago.
* Have had a blood transfusion or severe blood loss within 3 months prior to screening, or have known hemoglobinopathy, hemolytic anemia or sickle cell anemia, or any other traits of hemoglobin abnormalities known to interfere with HbA1c methodology.
* Are receiving chronic (lasting longer than 14 consecutive days) systemic glucocorticoid therapy (excluding topical, intra-articular, intraocular and inhaled prescriptions), or have received such therapy within the 4 weeks immediately preceding screening.
* Have an irregular sleep/wake cycle (for example, patients who sleep during the day and work during the night), in the investigator's opinion.
* Have known hypersensitivity or allergy to any of the study insulins or their excipients.
* Are breastfeeding or pregnant, or intend to become pregnant during the course of the study, or are sexually active women of childbearing potential not actively practicing birth control by a method determined by the investigator to be medically acceptable.
* Are currently enrolled in, or discontinued within the last 30 days from, a clinical trial involving an off-label use of an investigational drug or device (other than the study drug/device used in this study), or concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study.
* Have previously completed or withdrawn from this study after having signed the informed consent document (ICD).
* Are unwilling or unable to comply with the use of a data collection device to directly record data from the patient.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2010-04; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9am - 5pm Eastern (UTC/GMT - 5hrs, EST), Study Director — Eli Lilly and Company
Locations (11):
- United States (11):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Concord, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aurora, Colorado
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hollywood, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., West Palm Beach, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Idaho Falls, Idaho
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Topeka, Kansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nashua, New Hampshire
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Albany, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Syracuse, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Asheville, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Austin, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Sequence A (L2D/L6D/A6D): Participants received Insulin Lispro 2D (L2D (Days)), Insulin Lispro 6D (L6D) and Insulin Aspart 6D (A6D) as per below dosing schedule Period 1: Lispro 2D, Period 2: Lispro 6D and Period 3: Insulin Aspart 6D
- Sequence B (L2D/A6D/L6D): Participants received Insulin Lispro 2D, Insulin Lispro 6D and Insulin Aspart 6D as per below dosing schedule Period 1:
  Insulin Lispro 2D, Period 2: Insulin Aspart 6D and Period 3: Insulin Lispro 6D.
- Sequence C (L6D/L2D/A6D): Participants received Insulin Lispro 2D, Insulin Lispro 6D and Insulin Aspart 6D as per below dosing schedule Period 1: Insulin Lispro 6D, Period 2: Insulin Lispro 2D and Period 3: Insulin Aspart 6D.
- Sequence D (L6D/A6D/L2D): Participants received Insulin Lispro 2D, Insulin Lispro 6D and Insulin Aspart 6D as per below dosing schedule Period 1:
  Insulin Lispro 6D, Period 2: Insulin Aspart 6D and Period 3: Insulin Lispro 2D.
- Sequence E (A6D/L2D/L6D): Participants received Insulin Lispro 2D, Insulin Lispro 6D and Insulin Aspart 6D as per below dosing schedule Period 1: Insulin Aspart 6D, Period 2: Insulin Lispro 2D and Period 3: Insulin Lispro 6D.
- Sequence F (A6D/L6D/L2D): Participants received Insulin Lispro 2D, Insulin Lispro 6D and Insulin Aspart 6D as per below dosing schedule Period 1: Insulin Aspart 6D, Period 2: Insulin Lispro 6D and Period 3: Insulin Lispro 2D.
Period: Study Period 1
Arm/Group | Sequence A (L2D/L6D/A6D) | Sequence B (L2D/A6D/L6D) | Sequence C (L6D/L2D/A6D) | Sequence D (L6D/A6D/L2D) | Sequence E (A6D/L2D/L6D) | Sequence F (A6D/L6D/L2D)
Started | 22 | 22 | 22 | 22 | 22 | 22
Received at Least One Dose of Study Drug | 22 | 22 | 22 | 22 | 22 | 20
Completed | 22 | 22 | 19 | 21 | 20 | 20
Not Completed | 0 | 0 | 3 | 1 | 2 | 2
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 2 | 0
Not completed — Sponsor Decision | 0 | 0 | 0 | 0 | 0 | 2
Period: Study Period 2
Arm/Group | Sequence A (L2D/L6D/A6D) | Sequence B (L2D/A6D/L6D) | Sequence C (L6D/L2D/A6D) | Sequence D (L6D/A6D/L2D) | Sequence E (A6D/L2D/L6D) | Sequence F (A6D/L6D/L2D)
Started | 22 | 22 | 19 | 21 | 20 | 20
Completed | 21 | 21 | 18 | 20 | 20 | 19
Not Completed | 1 | 1 | 1 | 1 | 0 | 1
Not completed — Entry Criteria Not Met | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 1
Period: Study Period 3
Arm/Group | Sequence A (L2D/L6D/A6D) | Sequence B (L2D/A6D/L6D) | Sequence C (L6D/L2D/A6D) | Sequence D (L6D/A6D/L2D) | Sequence E (A6D/L2D/L6D) | Sequence F (A6D/L6D/L2D)
Started | 21 | 21 | 18 | 20 | 20 | 19
Completed | 20 | 21 | 18 | 20 | 18 | 19
Not Completed | 1 | 0 | 0 | 0 | 2 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Sequence A (L2D/L6D/A6D): Participants received Insulin Lispro 2D (2 Days), Insulin Lispro 6D and Insulin Aspart 6D as per below dosing schedule Period 1: Lispro 2D, Period 2: Lispro 6D and Period 3: Insulin Aspart 6D.
- Total: Total of all reporting groups
Arm/Group | Sequence A (L2D/L6D/A6D) | Sequence B (L2D/A6D/L6D) | Sequence C (L6D/L2D/A6D) | Sequence D (L6D/A6D/L2D) | Sequence E (A6D/L2D/L6D) | Sequence F (A6D/L6D/L2D) | Total
Number analyzed (Participants) | 22 | 22 | 22 | 22 | 22 | 22 | 132
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.28 (19.62) | 36.61 (14.07) | 42.63 (17.39) | 47.23 (18.78) | 41.15 (14.22) | 38.34 (14.93) | 41.37 (16.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 16 | 15 | 14 | 18 | 18 | 96
  Male | 7 | 6 | 7 | 8 | 4 | 4 | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 4 | 1 | 0 | 3 | 3 | 12
  Not Hispanic or Latino | 21 | 18 | 21 | 22 | 19 | 19 | 120
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 0 | 0 | 0 | 1
  White | 22 | 21 | 22 | 21 | 22 | 21 | 129
  More than one race | 0 | 0 | 0 | 1 | 0 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 22 | 22 | 22 | 22 | 22 | 22 | 132

OUTCOME MEASURES:

1. Primary Outcome: Mean of Last Five 7-point Self Monitored Blood Glucose (SMBG) Taken on Day 6 for Insulin Lispro 6D and Day 2 for Insulin Lispro 2D and Day 6 for Insulin Aspart 6D Pump Reservoir In-use
Time Frame: 8 weeks of each treatment
Population: All randomized participants who completed at least one post-randomization visit. Those included in the Primary analysis had to have at least one reservoir in-use cycle with an SMBG measurement on Day 6 during the pre-specified collection period.
Measure: Mean (Standard Deviation); unit: millimoles per liter (mmol/L)
Groups:
- Insulin Lispro 2 Day: Insulin Lispro 2 Day (L2D) administered by infusion pump for 8 week treatment period.
- Insulin Lispro 6 Day: Insulin Lispro 6 Day (L6D) administered by infusion pump for 8 weeks.
- Insulin Aspart 6 Day: Insulin Aspart 6 Day (A6D) administered by infusion pump for 8 weeks.
Arm/Group | Insulin Lispro 2 Day | Insulin Lispro 6 Day | Insulin Aspart 6 Day
Number analyzed (Participants) | 119 | 116 | 117
millimoles per liter (mmol/L) | 9.03 (2.17) | 9.33 (2.31) | 8.72 (1.82)
Statistical Analysis 1: Comparison: Insulin Lispro 6 Day vs Insulin Aspart 6 Day; This was the primary gated analysis; Test type: Non-Inferiority or Equivalence — Non-inferiority margin of 0.6 mmol/L was used; Least Squares Mean Difference = 0.48, 95% CI 2-sided [0.20 to 0.76] — Least Squares Mean Difference = Insulin Lispro 6 Day minus Insulin Aspart 6 Day; adjusted for Treatment + Sequence + Period + Age stratum + Baseline HbA1c

2. Secondary Outcome: Mean SMBG
Description: Mean SMBG for combined periods; all reported SMBG values on days 1-6 for Insulin Lispro 6 Day and Insulin Aspart 6 Day, and days 1-2 for Insulin Lispro 2 Day.
Time Frame: 8 weeks for each treatment
Population: All randomized participants who completed at least one post-randomization visit and one SMBG measurement on Day 2 for insulin lispro 2 day or Day 6 for the respective treatment arm: insulin lispro 6 day and insulin aspart 6 day.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Insulin Lispro 2 Day | Insulin Lispro 6 Day | Insulin Aspart 6 Day
Number analyzed (Participants) | 122 | 122 | 122
mmol/L | 8.79 (2.73) | 9.01 (2.87) | 8.83 (2.71)
Statistical Analysis 1: Comparison: Insulin Lispro 6 Day vs Insulin Aspart 6 Day; Test type: Non-Inferiority or Equivalence — Non-inferiority margin of 0.6 mmol/L was used; Least Squares Mean Difference = 0.22, 95% CI 2-sided [-0.07 to 0.52] — Least Squares Mean Difference = Insulin Lispro 6 Day minus Insulin Aspart 6 Day; adjusted for Treatment + Sequence + Period + Age Stratum + Baseline HbA1c; where participant is treated as a random effect
Statistical Analysis 2: Comparison: Insulin Lispro 2 Day vs Insulin Lispro 6 Day; Test type: Non-Inferiority or Equivalence — Non-inferiority margin of 0.6 mmol/L was used; Least Squares Mean Difference = 0.25, 95% CI 2-sided [-0.05 to 0.56] — [estimate comment as in outcome 2, analysis 1]

3. Secondary Outcome: Mean Daily Insulin Dose (Total, Basal, and Bolus)
Time Frame: 8 weeks for each treatment
Population: All randomized participants who completed at least one post-randomization visit. Participants included in insulin analyses are only those for whom data existed regarding insulin dose.
Measure: Mean (Standard Deviation); unit: Units (U) of insulin
Arm/Group | Insulin Lispro 2 Day | Insulin Lispro 6 Day | Insulin Aspart 6 Day
Number analyzed (Participants) | 117 | 117 | 117
Units (U) of insulin
  Daily Bolus Insulin: number analyzed (Participants) | 116 | 115 | 115
  Daily Bolus Insulin | 14.33 (5.88) | 14.51 (6.33) | 14.44 (6.11)
  Daily Basal Insulin | 18.62 (9.32) | 18.77 (8.89) | 18.34 (8.72)
  Daily Total Insulin | 32.36 (10.28) | 32.37 (10.12) | 31.99 (10.15)
Statistical Analysis 1: Comparison: Insulin Lispro 6 Day vs Insulin Aspart 6 Day; Test type: Superiority or Other; Least Squares Mean Difference = 0.11, 95% CI 2-sided [-0.29 to 0.51] — Least Squares Mean Difference of Daily Bolus Insulin = Insulin Lispro 6 Day minus Insulin Aspart 6 Day; adjusted for Treatment + Sequence + Period + Baseline Insulin Basal/Bolus/Total Dose + Age Stratum
Statistical Analysis 2: Comparison: Insulin Lispro 2 Day vs Insulin Lispro 6 Day; Test type: Superiority or Other; Least Squares Mean Difference = 0.16, 95% CI 2-sided [-0.41 to 0.73] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: Insulin Lispro 6 Day vs Insulin Aspart 6 Day; Test type: Superiority or Other; Least Squares Mean Difference = 0.03, 95% CI 2-sided [-0.18 to 0.24] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 4: Comparison: Insulin Lispro 2 Day vs Insulin Lispro 6 Day; Test type: Superiority or Other; Least Squares Mean Difference = -0.14, 95% CI 2-sided [-0.56 to 0.27] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 5: Comparison: Insulin Lispro 6 Day vs Insulin Aspart 6 Day; Test type: Superiority or Other; Least Squares Mean Difference = 0.06, 95% CI 2-sided [-0.48 to 0.60] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 6: Comparison: Insulin Lispro 2 Day vs Insulin Lispro 6 Day; Test type: Superiority or Other; Least Squares Mean Difference = -0.10, 95% CI 2-sided [-0.85 to 0.65] — [estimate comment as in outcome 3, analysis 1]

4. Secondary Outcome: Change From Baseline to 8 Weeks Endpoint for Each Treatment in Hemoglobin A1c (HbA1c) Values
Time Frame: Baseline, 8 weeks for each treatment
Population: All randomized participants who completed at least one post-randomization visit, and had a baseline and a post-randomization HbA1c measurement for the respective treatment period. Last Observation Carried Forward (LOCF) method was utilized in this analysis.
Measure: Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin
Arm/Group | Insulin Lispro 2 Day | Insulin Lispro 6 Day | Insulin Aspart 6 Day
Number analyzed (Participants) | 121 | 120 | 121
percentage of glycosylated hemoglobin | -0.04 (0.59) | 0.06 (0.56) | 0.00 (0.53)
Statistical Analysis 1: Comparison: Insulin Lispro 6 Day vs Insulin Aspart 6 Day; Test type: Superiority or Other; Least Squares Mean Difference = 0.06, 95% CI 2-sided [-0.02 to 0.14] — Least Squares Mean Difference = Insulin Lispro 6 Day minus Insulin Aspart 6 Day; adjusted for Treatment + Period + Sequence + Baseline HbA1c
Statistical Analysis 2: Comparison: Insulin Lispro 2 Day vs Insulin Lispro 6 Day; Test type: Superiority or Other; Least Squares Mean Difference = 0.09, 95% CI 2-sided [0.01 to 0.18] — [estimate comment as in outcome 4, analysis 1]

5. Secondary Outcome: Number of Participants Who Achieve or Maintain an HbA1c Less Than or Equal to 6.5% and Less Than 7%
Time Frame: 8 weeks for each treatment
Population: All randomized participants who completed a post-randomization visit and had an HbA1c measurement for the respective treatment period.
Measure: Number; unit: participants
Arm/Group | Insulin Lispro 2 Day | Insulin Lispro 6 Day | Insulin Aspart 6 Day
Number analyzed (Participants) | 121 | 120 | 121
participants
  HbA1c ≤6.5% | 21 | 16 | 18
  HbA1c <7% | 40 | 38 | 44
Statistical Analysis 1: Comparison: Insulin Lispro 6 Day vs Insulin Aspart 6 Day; Test type: Superiority or Other; Odds Ratio (OR) = 0.93, 95% CI 2-sided [0.50 to 1.75] — Odds Ratio of HbA1c ≤6.5% for Insulin Lispro 6 Day versus Insulin Aspart 6 Day
Statistical Analysis 2: Comparison: Insulin Lispro 2 Day vs Insulin Lispro 6 Day; Test type: Superiority or Other; Odds Ratio (OR) = 0.69, 95% CI 2-sided [0.29 to 1.67] — Odds Ratio of HbA1c ≤6.5% for Insulin Lispro 6 Day versus Insulin Lispro 2 Day
Statistical Analysis 3: Comparison: Insulin Lispro 6 Day vs Insulin Aspart 6 Day; Test type: Superiority or Other; Odds Ratio (OR) = 0.89, 95% CI 2-sided [0.56 to 1.41] — Odds Ratio of HbA1c <7% for Insulin Lispro 6 Day versus Insulin Aspart 6 Day
Statistical Analysis 4: Comparison: Insulin Lispro 2 Day vs Insulin Lispro 6 Day; Test type: Superiority or Other; Odds Ratio (OR) = 1.04, 95% CI 2-sided [0.66 to 1.64] — Odds Ratio of HbA1c <7% for Insulin Lispro 6 Day versus Insulin Lispro 2 Day

6. Secondary Outcome: Percentage of Participants With Hyperglycemia
Description: Hyperglycemia was defined as an event with (1) a measured blood glucose concentration >250 milligrams per deciliter (mg/dL) (13.9 mmol/L) and ≥3 hours after eating, or (2) a measured blood glucose concentration >300 mg/dL (16.7 mmol/L) and <3 hours after eating.
Time Frame: 8 weeks for each treatment
Population: All randomized participants who received at least one dose of study drug. Participants included in hyperglycemia analyses are only those for whom data existed regarding hyperglycemia.
Measure: Number; unit: percentage of participants
Arm/Group | Insulin Lispro 2 Day | Insulin Lispro 6 Day | Insulin Aspart 6 Day
Number analyzed (Participants) | 122 | 127 | 124
percentage of participants | 99.2 | 98.4 | 98.4
Statistical Analysis 1: Comparison: Insulin Lispro 6 Day vs Insulin Aspart 6 Day; Test type: Superiority or Other; p = 1.00, Gart's Test — P-value computed using Treatment comparison Gart's Test. Participants represented in both treatment groups and with non-missing incidence value in each treatment period are used for p-value calculation

7. Secondary Outcome: Hyperglycemic Episode Rate Per 30 Days
Description: Hyperglycemia was defined as an episode with (1) a measured blood glucose concentration >250 milligrams per deciliter (mg/dL) (13.9 mmol/L) and ≥3 hours after eating, or (2) a measured blood glucose concentration >300 mg/dL (16.7 mmol/L) and <3 hours after eating. Rate is presented as the number of hyperglycemic episodes adjusted for 30 days.
Time Frame: 8 weeks for each treatment
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: hyperglycemic episodes per 30 days
Arm/Group | Insulin Lispro 2 Day | Insulin Lispro 6 Day | Insulin Aspart 6 Day
Number analyzed (Participants) | 122 | 127 | 124
hyperglycemic episodes per 30 days | 15.91 (12.78) | 16.91 (13.98) | 15.76 (12.04)
Statistical Analysis 1: Comparison: Insulin Lispro 6 Day vs Insulin Aspart 6 Day; Test type: Superiority or Other; p = 0.164, Negative Binomial Test — P-value computed using a negative binomial test including factors for treatment, period, and sequence
Statistical Analysis 2: Comparison: Insulin Lispro 2 Day vs Insulin Lispro 6 Day; Test type: Superiority or Other; p = 0.185, Negative Binomial Test — P-value computed using a negative binomial test including factors for treatment, period, and sequence

8. Secondary Outcome: Percentage of Participants With Pump Complications
Description: Overall Pump Complications were any combination of: tubing clogged, kinked, disconnected, pulled out, blood in tubing; too much heat, too much cold, empty reservoir, low battery, occlusion alarm, no delivery alarm; at site - skin abscess, excessive redness, swelling (not nodule), bleeding, bruising; reservoir change (infusion set change reason only); and other. When either a reservoir change or an infusion set change was reported, participants were questioned whether change was early (prior to 6 days for L6D or A6D, or prior to 2 days for L2D). If 'yes', then recorded as premature change.
Time Frame: 8 weeks for each treatment
Population: All randomized participants who completed at least one post-randomization visit. Participants included in pump complication analyses are only those for whom data existed regarding pump complications.
Measure: Number; unit: percentage of participants
Arm/Group | Insulin Lispro 2 Day | Insulin Lispro 6 Day | Insulin Aspart 6 Day
Number analyzed (Participants) | 122 | 127 | 124
percentage of participants
  Pump Complication: Premature Reservoir Change | 23.8 | 38.6 | 36.3
  Pump Complication: Premature Infusion Set Change | 42.6 | 59.1 | 56.5
Statistical Analysis 1: Comparison: Insulin Lispro 6 Day vs Insulin Aspart 6 Day; Test type: Superiority or Other; p = 0.736, Gart's Test — P-value for Premature Reservoir Change. P-value computed using Treatment comparison Gart's Test. Participants represented in both treatment groups and with non-missing incidence value in each treatment period are used for p-value calculation
Statistical Analysis 2: Comparison: Insulin Lispro 2 Day vs Insulin Lispro 6 Day; Test type: Superiority or Other; p = 0.006, Gart's Test — [p-value comment as in outcome 8, analysis 1]
Statistical Analysis 3: Comparison: Insulin Lispro 6 Day vs Insulin Aspart 6 Day; Test type: Superiority or Other; p = 1.00, Gart's Test — P-value for Premature Infusion Set Change. P-value computed using Treatment comparison Gart's Test. Participants represented in both treatment groups and with non-missing incidence value in each treatment period are used for p-value calculation
Statistical Analysis 4: Comparison: Insulin Lispro 2 Day vs Insulin Lispro 6 Day; Test type: Superiority or Other; p = 0.017, Gart's Test — [p-value comment as in outcome 8, analysis 3]

9. Secondary Outcome: Pump Complication Rate Per 30 Days
Description: as for outcome 8
Time Frame: 8 weeks for each treatment
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: pump complications per 30 days
Arm/Group | Insulin Lispro 2 Day | Insulin Lispro 6 Day | Insulin Aspart 6 Day
Number analyzed (Participants) | 122 | 127 | 124
pump complications per 30 days
  Pump Complication: Premature Reservoir Change | 0.16 (0.34) | 0.40 (0.76) | 0.51 (1.05)
  Pump Complication: Premature Infusion Set Change | 0.44 (0.65) | 0.84 (1.18) | 0.94 (1.35)
Statistical Analysis 1: Comparison: Insulin Lispro 6 Day vs Insulin Aspart 6 Day; Test type: Superiority or Other; p = 0.471, Negative Binomial Test — P-value for Premature Reservoir Change. P-value is computed using negative binomial test including factors for treatment, period and sequence
Statistical Analysis 2: Comparison: Insulin Lispro 2 Day vs Insulin Lispro 6 Day; Test type: Superiority or Other; p < 0.001, Negative Binomial Test — [p-value comment as in outcome 9, analysis 1]
Statistical Analysis 3: Comparison: Insulin Lispro 6 Day vs Insulin Aspart 6 Day; Test type: Superiority or Other; p = 0.737, Negative Binomial Test — P-value for Premature Infusion Set Change. P-value is computed using negative binomial test including factors for treatment, period and sequence
Statistical Analysis 4: Comparison: Insulin Lispro 2 Day vs Insulin Lispro 6 Day; Test type: Superiority or Other; p < 0.001, Negative Binomial Test — [p-value comment as in outcome 9, analysis 3]

10. Secondary Outcome: Percentage of Participants With Hypoglycemia
Description: Hypoglycemia was defined as an event which was associated with
  1. reported signs and symptoms of hypoglycemia, and/or
  2. a documented blood glucose (BG) concentration of ≤ 70 mg/dL (3.9 mmol/L).
Time Frame: 8 weeks for each treatment
Population: All randomized participants who received at least one dose of study drug. Participants included in hypoglycemia analyses are only those for whom data existed regarding hypoglycemia.
Measure: Number; unit: percentage of participants
Arm/Group | Insulin Lispro 2 Day | Insulin Lispro 6 Day | Insulin Aspart 6 Day
Number analyzed (Participants) | 122 | 127 | 124
percentage of participants | 100.0 | 100.0 | 99.2

11. Secondary Outcome: Hypoglycemia Episode Rate Per 30 Days
Description: Hypoglycemia was defined as an event which was associated with
  1. reported signs and symptoms of hypoglycemia, and/or
  2. a documented blood glucose (BG) concentration of ≤ 70 mg/dL (3.9 mmol/L). Rate is presented as the number of hypoglycemic episodes adjusted for 30 days.
Time Frame: 8 weeks for each treatment
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: hypoglycemic episodes per 30 days
Arm/Group | Insulin Lispro 2 Day | Insulin Lispro 6 Day | Insulin Aspart 6 Day
Number analyzed (Participants) | 122 | 127 | 124
hypoglycemic episodes per 30 days | 17.90 (11.13) | 15.66 (12.29) | 17.52 (11.76)
Statistical Analysis 1: Comparison: Insulin Lispro 6 Day vs Insulin Aspart 6 Day; Test type: Superiority or Other; p = 0.006, Negative Binomial Test — P-value is computed using negative binomial test including factors for treatment, period and sequence
Statistical Analysis 2: Comparison: Insulin Lispro 2 Day vs Insulin Lispro 6 Day; Test type: Superiority or Other; p = 0.002, Negative Binomial Test — P-value is computed using negative binomial test including factors for treatment, period and sequence

12. Secondary Outcome: Change From Baseline to 8 Weeks Endpoint for Each Treatment in Weight
Time Frame: Baseline, 8 weeks for each treatment
Population: All randomized participants who received at least one dose of study drug and had both baseline and post-baseline weight measurements for the respective treatment period.
Measure: Mean (Standard Deviation); unit: kilograms (kg)
Arm/Group | Insulin Lispro 2 Day | Insulin Lispro 6 Day | Insulin Aspart 6 Day
Number analyzed (Participants) | 121 | 122 | 122
kilograms (kg) | 0.44 (2.13) | 0.34 (2.04) | 0.65 (2.13)
Statistical Analysis 1: Comparison: Insulin Lispro 6 Day vs Insulin Aspart 6 Day; Test type: Superiority or Other; p = 0.060, Crossover Model — P-value computed using crossover model. Response = Treatment + Sequence + Period + Age stratum + Baseline Body Weight
Statistical Analysis 2: Comparison: Insulin Lispro 2 Day vs Insulin Lispro 6 Day; Test type: Superiority or Other; p = 0.486, Crossover Model — P-value computed using crossover model. Response = Treatment + Sequence + Period + Age stratum + Baseline Body Weight

13. Secondary Outcome: Change From Baseline to 8 Weeks Endpoint for Each Treatment in Blood Pressure
Time Frame: Baseline, 8 weeks for each treatment
Population: All randomized participants who received at least one dose of study drug and had both baseline and post-baseline blood pressure measurements for the respective treatment period.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Insulin Lispro 2 Day | Insulin Lispro 6 Day | Insulin Aspart 6 Day
Number analyzed (Participants) | 121 | 122 | 123
mmHg
  Systolic Blood Pressure (SBP) | 0.80 (12.82) | 0.80 (12.52) | -1.07 (12.06)
  Diastolic Blood Pressure (DBP) | -0.14 (8.24) | 1.37 (7.62) | -0.33 (7.88)
Statistical Analysis 1: Comparison: Insulin Lispro 6 Day vs Insulin Aspart 6 Day; Test type: Superiority or Other; p = 0.056, Crossover Model — P-value is for Systolic Blood Pressure. P-value computed using crossover model. Response = Treatment + Sequence + Period + Age stratum + Baseline Systolic Blood Pressure
Statistical Analysis 2: Comparison: Insulin Lispro 2 Day vs Insulin Lispro 6 Day; Test type: Superiority or Other; p = 0.805, Crossover Model — [p-value comment as in outcome 13, analysis 1]
Statistical Analysis 3: Comparison: Insulin Lispro 6 Day vs Insulin Aspart 6 Day; Test type: Superiority or Other; p = 0.020, Crossover Model — P-value is for Diastolic Blood Pressure. P-value computed using crossover model. Response = Treatment + Sequence + Period + Age stratum + Baseline Diastolic Blood Pressure
Statistical Analysis 4: Comparison: Insulin Lispro 2 Day vs Insulin Lispro 6 Day; Test type: Superiority or Other; p = 0.051, Crossover Model — [p-value comment as in outcome 13, analysis 3]

ADVERSE EVENTS:
Time Frame: Up To 8 weeks
Description: There are gender specific adverse events, only occurring in male or female participants. The number of participants exposed has been adjusted accordingly.
Arm/Group | Insulin Lispro 2 Day | Insulin Lispro 6 Day | Insulin Aspart 6 Day
Serious Adverse Events (participants affected / at risk) | 3/122 | 8/127 | 10/124
Other Adverse Events (participants affected / at risk) | 71/122 | 68/127 | 71/124
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Insulin Lispro 2 Day (N=122) | Insulin Lispro 6 Day (N=127) | Insulin Aspart 6 Day (N=124)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Sternal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 3 (4) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2) | 4 (5) | 9 (11) — These events were severe hypoglycemic events.
Cervical myelopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0/90 (0) | 0/93 (0) | 1/90 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Insulin Lispro 2 Day (N=122) | Insulin Lispro 6 Day (N=127) | Insulin Aspart 6 Day (N=124)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 4 (4) | 3 (3) | 4 (4)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 5 (5) | 2 (2) | 4 (4)
Asthenia (General disorders) | 0 (0) | 2 (2) | 1 (1)
Chills (General disorders) | 2 (2) | 0 (0) | 1 (1)
Infusion site erythema (General disorders) | 1 (1) | 1 (1) | 2 (2)
Infusion site haemorrhage (General disorders) | 1 (1) | 1 (1) | 2 (3)
Infusion site mass (General disorders) | 1 (1) | 1 (1) | 2 (2)
Pyrexia (General disorders) | 2 (2) | 5 (5) | 2 (2)
Ear infection (Infections and infestations) | 1 (1) | 3 (3) | 1 (1)
Fungal infection (Infections and infestations) | 2 (3) | 2 (2) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 5 (5) | 2 (2) | 3 (3)
Influenza (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
Nasopharyngitis (Infections and infestations) | 10 (11) | 11 (12) | 13 (14)
Pharyngitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Sinusitis (Infections and infestations) | 4 (4) | 1 (1) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 10 (10) | 6 (6) | 9 (10)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (2) | 3 (4)
Viral infection (Infections and infestations) | 1 (1) | 2 (2) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 1 (1)
Urine ketone body present (Investigations) | 0 (0) | 1 (1) | 2 (3)
Hyperlipidaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 2 (2)
Tendonitis (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 3 (3)
Headache (Nervous system disorders) | 6 (7) | 3 (3) | 3 (3)
Depression (Psychiatric disorders) | 2 (2) | 2 (2) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (3) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 4 (4) | 5 (5)
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1)
Rhinitis seasonal (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 2 (2)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4) | 3 (3)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Subcutaneous nodule (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 2 (2)
Vulvovaginal Mycotic Infection (Infections and infestations) | 0/90 (0) | 0/93 (0) | 1/90 (1)
Smear Cervix Abnormal (Infections and infestations) | 0/90 (0) | 1/93 (1) | 0/90 (0)

LIMITATIONS AND CAVEATS:
Input to primary endpoint measurements (SMBG) contained approximately 40% missing data. Several analyses to account for missing data have been conducted and results from these additional analyses were consistent with results of original analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days